CLINICAL TRIAL: NCT02841943
Title: Fluid Responsiveness After Cardiac Surgery (FRACAS) Study
Brief Title: Fluid Responsiveness After CArdiac Surgery Study
Acronym: FRACAS
Status: Completed | Type: Observational
Sponsor: South West Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Anders Aneman, Senior Staff Specialist, South West Sydney Local Health District
Other Study IDs: LIVICU001
Record Dates: First submitted 2016-07-15; First posted 2016-07-22 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Critically Ill; Hypovolemia
Keywords: Fluid responsiveness; Near-infrared spectroscopy; Thoracic surgery; Hypovolemia; veno-arterial carbon dioxide gradient; arterio-venous oxygen gradient; hypercarbia; Carotid artery; ultrasonography; Doppler
MeSH Terms: conditions — Critical Illness; Hypovolemia; Hypercapnia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Study Design: Prospective observational study

Study Location: Liverpool Hospital Intensive Care Unit, South Western Sydney Local Health District, Sydney, Australia.

Target study size: 100 patients

Ethics: Approved by the local Human Research and Ethics Council (HREC) at Liverpool Hospital (LPOOL) as a Low Negligible Risk (LNR) project [HREC/LNR/14/LPOOL/295, HREC/LNR/15/LPOOL47, HREC/LNR/14/LPOOL/150]

Participants: Post cardiac surgical patients admitted to the Intensive Care Unit between March-October 2016

Aims:

1. to determine the descriptive and predictive value of variables (outlined below) related to oxygen delivery/consumption in regards to the effects of intravascular volume expansion
2. to assess correlations between central and peripheral variables (outlined below) relevant to oxygen delivery/consumption
3. to assess correlations between a set of variables (outline below) and patient centred outcomes in ICU and in hospital

Main variables collected:

1. Tissue oxygen saturation by peripheral Near-Infrared Spectroscopy (NIRS)
2. Common carotid arterial Doppler
3. Arterial/mixed venous/central venous blood gas analyses
4. Haemodynamic parameters
5. Organ support measures

Data collection time points:

1. ICU admission (within 30 minutes)
2. Before administration of a fluid bolus
3. After administration of a fluid bolus
4. 6 hours after ICU admission
5. Morning of first postoperative day (12-24 hours)

Outcome measures:

1. the response to intravascular volume expansion
2. ICU mortality, morbidity and length of stay and hospital mortality and length of stay

Data analysis:

1. Clinical data are collected bedside using an electronic case record form
2. Descriptive statistics
3. Paired and unpaired comparative
4. Correlative and predictive statistics

DETAILED DESCRIPTION:
This prospective observational study program has a set of objectives within three major domains that will be analysed separately and synergistically:

Peripheral near infra-red spectroscopy (NIRS)

Aims:

1. to describe the effects of non-sanguineous intravascular volume expansion on systemic oxygen delivery
2. to describe how changes in systemic oxygen delivery impact on peripheral oxygen kinetics as measured by tissue oxygen saturation (StO2) in the thenar and forearm regions at rest and using a vascular occlusion test
3. to determine the clinical applicability of using thenar and forearm NIRS to guide haemodynamic optimisation following cardiac surgery
4. to assess the relation between systemic and peripheral oxygen kinetics vs. onset of organ dysfunction and need for extended stay in ICU following cardiac surgery

Hypotheses:

1. Peripheral oxygen kinetics using NIRS offer more specific guidance for haemodynamic optimisation post cardiac surgery compared to using systemic variables only
2. Impaired peripheral oxygen kinetics as assessed using NIRS can be used to identify patients at risk for developing organ dysfunction or needing extended period of ICU support an earlier stage compared to traditional systemic variables

Main measurements:

1. peripheral near infrared spectroscopy (NIRS) measuring tissue oxygen saturation (StO2) at the thenar eminence and forearm during a 3 minute vascular occlusion test at 50mmHg above systolic pressure, following the establishment of a baseline (an StO2 average over 3 minutes with less than 5% variability)
2. StO2 measurements are repeated at 30 minutes intervals during the first 6 hours following admission to ICU.
3. vascular occlusion tests are repeated before and after volume expansion.

Cardiac output and common carotid Doppler sonography

Aims:

1. to apply computerised algorithms to derive advanced haemodynamic information (mean systemic filling pressure, heart efficiency, vascular compliance) in patients requiring fluid boluses following cardiac surgery
2. to correlate changes in cardiac output, cardiac power and estimates of fluid responsiveness using the pulmonary artery catheter with the variables mean systemic filling pressure and heart efficiency
3. to characterise indices of fluid responsiveness by measuring volume efficiency
4. to determine the impact of changes in vascular resistance state on the assessment of changes in volume state in the post-operative cardiac surgery period
5. to assess the relation between fluid responsiveness, fluid management and clinical outcomes in ICU following cardiac surgery
6. to evaluate the potential for carotid Doppler blood flow measurements as a surrogate parameter for cardiac output, including incorporation into computerised algorithms

Hypotheses:

1. the derived measures of mean systemic filling pressure and heart efficiency are superior to identify fluid responsiveness compared to cardiac output measurements alone in patients following cardiac surgery
2. carotid Doppler blood flow measurements can be used as a surrogate parameter for cardiac output and in particular for changes in cardiac output when fluid responsiveness is investigated

Main measurements:

1. Pulmonary arterial thermodilution studies (for cardiac output, stroke volume, cardiac index) by at least triplicate injections within a ± 10% range
2. Computerised algorithms are used to derive an analogue mean systemic filling pressure, heart efficiency, volume efficiency based on cardiac output, central venous pressure and mean arterial pressure
3. Common carotid Doppler sonography to measure vessel diameter, cross sectional area and time average mean velocity to generate blood flow as well as respirophasic peak flow velocity variation

Oxygen and carbon dioxide gradients

Aims:

1. to assess any insufficiency of oxygen delivery to match the oxygen consumption, resulting in anaerobic metabolism, by determining i) arteriovenous concentration gradients for lactate, ii) the venoarterial carbon dioxide tension gradient [P(v-a)CO2] and the arteriovenous oxygen content gradient ([C(a-v)O2]
2. to assess whether central venous blood gas analyses can substitute pulmonary arterial (mixed venous) blood gas analyses in the [P(v-a)CO2] and [C(a-v)O2] gradients and ratio
3. to assess whether arteriovenous O2 and CO2 gradients are more specific and contemporaneous measures of anaerobic metabolism compared to serum lactate

Hypotheses:

1. Changes in [C(a-v)O2] and [P(v-a)CO2] gradients can be used as prognostic markers with persistently abnormal values correlating with the presence and degree of organ failure
2. Changes in [C(a-v)O2] and [P(v-a)CO2] gradients can be used as targets during haemodynamic optimisation
3. Cumulative measurements of [C(a-v)O2] and [P(v-a)CO2] gradients to generate an area under the curve value can be used to assess and target the presence of an oxygen debt

Main measurements

1) Central venous, pulmonary arterial (mixed venous) and arterial blood gas analyses (pO2, pCO2, bicarbonate and lactate concentrations)

A fluid bolus will be administered as 250ml or 500ml of fluid (crystalloid or colloid) at 1500ml/hour. Measurements will be conducted immediately before fluid administration and 10 minutes post fluid cessation.

The following risk scores will be calculated: Sequential Organ Failure Assessment (SOFA), Acute Physiology and Chronic Health Evaluation (APACHE II and III), Simplified Acute Physiology Score (SAPS2), Australian New Zealand Risk of Death (ANZROD), Euroscore 2.

Routine biochemical tests will be recorded including electrolytes, renal function tests, liver function tests.

ELIGIBILITY:
Inclusion Criteria:

* Admitted following elective cardiac surgery
* Adult (>18 years of age)
* Pulmonary artery, central venous and arterial catheters inserted

Exclusion Criteria:

* Emergency Patients (surgery immediately or within 12 hours of admission to hospital)
* Children (< 18 years of age)
* Patients admitted to ICU with ongoing extracorporeal circulatory support
* Patients re-admitted to ICU within same index hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients electively admitted to the Intensive Care Unit following cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2016-03; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Fluid bolus responsiveness | Approximately 30 minutes
  Fluid responsiveness will be determined by any increase in cardiac output (continuous outcome) or by a 10-15% increase in cardiac output (dichotomous outcome) following bolus volume expansion
Volume management responsiveness | Approximately 6 hours
  Responders will be defined as patients with an improvement (change towards normal physiological values) following cumulative volume expansion in any variable(s) used to assess oxygen delivery/consumption balance

SECONDARY OUTCOMES:
Morbidity | At ICU discharge, an average of 4 days
  Use and extent of measures to support organ function such as mechanical ventilation, mechanical and pharmacological cardiovascular interventions, renal replacement therapy whilst admitted to ICU as well as length of admission to ICU.
Mortality | Up to 3 months
  Vital status censored at discharge from ICU and hospital

CONTACTS AND LOCATIONS:
Overall Officials: Anders Aneman, MD, PhD, Study Director — Liverpool Hospital, South Western Sydney Local Health District
Locations (1):
- Intensive Care Unit, Liverpool Hospital, South Western Sydney Local Health District, Liverpool, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta K, Sondergaard S, Parkin G, Leaning M, Aneman A. Applying mean systemic filling pressure to assess the response to fluid boluses in cardiac post-surgical patients. Intensive Care Med. 2015 Feb;41(2):265-72. doi: 10.1007/s00134-014-3611-2. Epub 2015 Jan 8. PMID 25567379
- [Background] Sondergaard S, Parkin G, Aneman A. Central venous pressure: soon an outcome-associated matter. Curr Opin Anaesthesiol. 2016 Apr;29(2):179-85. doi: 10.1097/ACO.0000000000000305. PMID 26825283
- [Background] Rangappa R, Sondergaard S, Aneman A. Improved consistency in interpretation and management of cardiovascular variables by intensive care staff using a computerised decision-support system. Crit Care Resusc. 2014 Mar;16(1):48-53. PMID 24588436